CLINICAL TRIAL: NCT06424197
Title: Colorectal Screening Fear-reduction and Racially-targeted Norm Messaging Entreaties to Increase Colorectal Cancer Screening Rates Among African Americans
Brief Title: Colorectal Cancer Screening Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oakland University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: IRB-FY2023-3; R21MD016506 (NIH)
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectcal Cancer Screening Targeted Message Intervention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Norm Based Messages (Experimental): One of 3 messaging entreaties based on normative perceptions of colorectal cancer screening, and one no norm-based messaging arm.
  Interventions: Other: Racial group-targeted messages
- Fear Reduction Message (Experimental): Participants randomized to receive (or not receive) messaging entreaty to address colorectal cancer screening fears.
  Interventions: Other: Racial group-targeted messages
- Commitment (Experimental): Participants randomized to indicate explicit commitment to return FIT Kits for processing.
  Interventions: Other: Explicit Commitment
- Control (No Intervention): Participants receive no health messages.

INTERVENTIONS:
Other: Racial group-targeted messages — Colorectal cancer screening messages targeted towards participants racial group.
  Arms: Fear Reduction Message; Norm Based Messages
Other: Explicit Commitment — Indicate explicit commitment to return at home screening kit.
  Arms: Commitment

SUMMARY:
Colorectal cancer (CRC) is one of the leading causes of cancer mortality in the United States, and African Americans (AfAms) still fare worse in CRC incidence and mortality compared to European Americans (EuAms). We propose to examine whether combining both fear-reduction and racially-targeted norm-based messages will increase at-home stool-based CRC screening receptivity and uptake for all African American regardless of level of racial identity. Given low return rates of at-home screening kits, we will also explore whether making an explicit commitment to return screening kits is associated with increased kit returns.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the leading causes of cancer mortality in the United States, and African Americans (AfAms) still fare worse in CRC incidence and mortality compared to European Americans (EuAms).Interventions to increase CRC screening rates among AfAms are instrumental to address the disparities in CRC incidence and mortality. Despite literature indicating that AfAms' fears (e.g., of colonoscopy procedures or cancer diagnosis) serve as barriers to CRC screening, no interventions have used theory-guided methods to directly target fear-based beliefs. Additionally, no research has examined the extent to which racial identity moderates the effects of racially targeted messaging, despite the ubiquity of using targeted health messaging entreaties among minority groups. This is particularly relevant given our work showing that racially-targeted screening entreaties increased CRC screening intentions among AfAms who identified less strongly, but depressed those intentions among AfAms who identified more strongly with their racial group. Lack of focus on other salient CRC screening barriers may have been off-putting to highly identified African Americans. We propose to examine whether combining both fear-reduction and racially-targeted norm-based messages will increase at-home stool-based CRC screening receptivity and uptake for all African American regardless of level of racial identity. Given low return rates of at-home screening kits, we will also explore whether making an explicit commitment to return screening kits is associated with increased kit returns.

Aim 1: To develop and refine a fear-reduction intervention guided by the theory of planned behavior and by published literature, in conjunction with AfAm community experts.

Aim 2: To examine whether the fear-reduction entreaty increases receptivity to, and uptake of at-home CRC screening when coupled with racially-targeted norm-based messages.

Aim 3: To examine the moderating roles of racial identity and perceived CRC risk on the effects of fear-reduction and racially-targeted norm-based messaging entreaties.

Aim 4: We will explore whether participants who make explicit commitments to return FIT Kits return them at a higher rate compared to those who do not make such commitments.

ELIGIBILITY:
Inclusion Criteria:

African American Overdue to colorectal cancer screening Has primary care physician Not at high risk for colorectal cancer

Exclusion Criteria:

Not meeting inclusion criteria

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
FIT Kit request | Immediately after survey
  FIT Kit request

SECONDARY OUTCOMES:
FIT Kit return | 3 months
  Mailing completed FIT Kit to lab for processing

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manning, PhD, Principal Investigator — Oakland University
Locations (1):
- Oakland University, Rochester, Michigan, United States

IPD SHARING:
Plan to Share IPD: No